CLINICAL TRIAL: NCT05672186
Title: Evaluating Diet, Food Insecurity, and Food Purchasing Outcomes of a Full-Service Mobile Food Market With a Cluster Randomized Trial
Brief Title: Mobile Food Market Cluster Randomized Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: social pro
Record Dates: First submitted 2022-12-12; First posted 2023-01-05 (Actual); Last update posted 2025-10-31 (Actual); Status verified 2025-10

CONDITIONS: Healthy Diet; Nutrition, Healthy

STUDY DESIGN:
Masking Description: Following site enrollment, sites will be randomized by wave to receive the full-service market intervention or serve as a waitlist control by the study statistician, who will be blinded to study site names. After randomization, the study statistician will be unblinded to site names by being given the key that matches sites with their assigned numbers. The study statistician will use this key to inform the mobile market co-investigator of site allocation to allow time for the mobile market to plan for market routes and schedules while baseline data collection is ongoing. Participants, site locations, the PI, university non-statistician trial investigators, and research staff will be blinded to site randomization results until baseline data collection is complete. Only the project manager and study statistician will be aware of the key (the link between the site names and the assigned site numbers linked to the data to be used in analysis) until analysis is complete.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Waitlist control (Sham Comparator): Participants in low-income neighborhoods and/or adjacent to low-income housing randomized to the control group will be placed on a waitlist to receive market service after follow- up data collection is complete.
  Interventions: Other: No intervention
- Experimental group (Experimental): Participants in low-income neighborhoods and/or adjacent to low-income housing randomized to the intervention group will receive the full-service market intervention following randomization.
  Interventions: Behavioral: Full-service market intervention

INTERVENTIONS:
Behavioral: Full-service market intervention — Full-service mobile market implementation: the market will visit intervention sites weekly. The market will carry items from all food groups including fresh, frozen and canned fruits and vegetables, whole grains, dairy/ dairy substitutes, proteins (e.g., frozen meat/fish, beans, eggs), and dry goods (e.g., cooking oil, spices). Prices on the market are affordable, approximately 10% lower than grocery stores.
  Arms: Experimental group
Other: No intervention — No intervention
  Arms: Waitlist control

SUMMARY:
Mobile food markets have been proposed as a strategy for mitigating health disparities related to poor nutrition and diet/weight-related health conditions because they bring low-cost, healthy food directly to underserved populations. Full-service mobile markets may improve multiple aspects of the diet by providing foods to meet all dietary needs through a convenient one-stop shop. The full-service mobile market to be tested (Twin Cities Mobile Market) sells nutritious and staple foods from a bus that regularly visits low-income neighborhoods. Foods are sold at prices ~10% below those of grocery stores. SNAP/EBT is accepted, and a state-funded fruit/vegetable incentive program (Market Bucks) is available to shoppers. Working in partnership with our community team members, we will enroll 12 total sites and recruit 22 participants per site (N=264). We will collect baseline data and randomize sites to either receive the full-service mobile market intervention or serve as the waitlist control. We will then implement the full-service mobile market at intervention sites, follow participants for 6 months, and collect follow-up data. After follow-up data collection, waitlist control sites will receive the full-service mobile market intervention. Diet quality will be assessed through dietary recall interviews, food insecurity will be assessed by survey, and fruit and vegetable purchases will be measured by collecting one month of food purchase tracking forms at baseline and follow-up data collection. Analyses will determine whether the full-service mobile market changes diet quality, food security, and food purchasing outcomes.

ELIGIBILITY:
Inclusion Criteria:

Community sites (e.g., public housing hi-rise, low-income senior living residence) must meet the following criteria:

* locale for low-income populations that experience difficulty in accessing healthy, affordable foods (e.g., public housing residences; low-income senior housing) or a community center in a low-income, low-food access (0.5 mile) census tract;
* willingness to be randomized to the intervention or waitlist control;
* located over 0.5 miles apart from other trial sites;
* willingness to allow for recruitment and data collection to occur in onsite community rooms

Participants must meet the following criteria:

* being aged 18 years or older;
* identifying as the primary food shopper in their household;
* being able to speak English or ASL;
* living within a half mile of the community site location; and
* reporting to be likely or somewhat likely to shop at the market in response to: "how likely would you be to shop regularly at the Twin Cities Mobile Market if it came to your neighborhood each week (response options: likely to unlikely).
* willing and able to participate in all study data collection activities

Exclusion Criteria:

* planning to move in the next 12 months
* currently shopping at the mobile market
* not having a phone number or mailing address
* presence of a condition or abnormality that would prohibit participation in the study or the quality of the data

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 262 (Actual)
Dates: Start 2023-01-12 (Actual); Primary Completion 2025-10-09 (Actual); Study Completion 2025-10-24 (Actual)

PRIMARY OUTCOMES:
Diet quality | At baseline and 6 month follow-up
  Trained research staff certified in collecting dietary recalls using Nutrition Data System for Research software will collect three 24-hour dietary recall interviews (2 weekdays, 1 weekend day) from each participant at each measurement period. Dietary recall data will be used to calculate the Health Eating Index Total Score.

SECONDARY OUTCOMES:
Food insecurity | At baseline and 6 month follow-up
  Food security in the past 6 months will be measured with the 18-item Household food security screening module of the USDA. From this measure, household food security status (food insecure or food secure) will be calculated per USDA guidelines for each time Food insecurity (yes, no) will be measured with the 18-item food security screening module of the USDA.
Level of food insecurity | At baseline and 6 month follow-up
  Food insecurity in the past 6 months will be measured with the 18-item food security screening module of the USDA. From this measure, household food security level (very low, low, marginal, and high food security) will be calculated per USDA guidelines for each time point, which will allow for calculation of level of food security prevalence at each time point.
Average weekly servings of fruits and vegetables procured | At baseline and 6 month follow-up
  Participants will use forms to record the fruits and vegetables they procured for their household and mail the forms to the researchers in prepaid addressed envelopes. Form data will be entered into Nutrition Data System for Research software to measure average weekly servings of fruits and vegetables procured.
Fruit and vegetables (servings/day) | At baseline and 6 month follow-up
  Trained research staff certified in collecting dietary recalls using Nutrition Data System for Research software will collect three 24-hour dietary recall interviews (2 weekdays, 1 weekend day) from each participant at each measurement period. Dietary recall data will be used to calculate the fruit and vegetables (servings/day) at baseline and follow-up.
Daily intake of energy (kcal/day) | At baseline and 6 month follow-up
  Trained research staff certified in collecting dietary recalls using Nutrition Data System for Research software will collect three 24-hour dietary recall interviews (2 weekdays, 1 weekend day) from each participant at each measurement period. Dietary recall data will be used to calculate the daily intake of energy (kcal/day).
Percent calories from added sugar | At baseline and 6 month follow-up
  Trained research staff certified in collecting dietary recalls using Nutrition Data System for Research software will collect three 24-hour dietary recall interviews (2 weekdays, 1 weekend day) from each participant at each measurement period. Dietary recall data will be used to calculate percent calories from added sugar.
Sodium (mg/day) | At baseline and 6 month follow-up
  Trained research staff certified in collecting dietary recalls using Nutrition Data System for Research software will collect three 24-hour dietary recall interviews (2 weekdays, 1 weekend day) from each participant at each measurement period. Dietary recall data will be used to calculate sodium (mg/day) intake.

CONTACTS AND LOCATIONS:
Overall Officials: Melissa Horning, PhD, RN, PHN, Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States

IPD SHARING:
Plan to Share IPD: Yes
The study protocol, statistical analysis plan, and consent form are available on the trial's clinicaltrials.gov registry (NCT05672186). Quarto (R Markdown) documents will describe and implement all data extraction, cleaning, and analysis steps, and the resulting files will be made publicly available alongside all publications resulting from this study. To support the reproducibility and replication of our findings, upon completion of the trial, we will share anonymized quantitative participant data used in publications of outcomes with the community partner and researchers. Proposals to access the data should be directed to horn0199@umn.edu.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: Upon completion of the trial
Access Criteria: Proposals to access the data should be directed to horn0199@umn.edu.

REFERENCES:
- [Derived] Horning ML, Gorman KS, Wagner S, Fulkerson JA, Wolfson J, Laska MN, Harnack L. Evaluating the impact of a full-service mobile food market on food security, diet quality and food purchases: a cluster randomised trial protocol and design paper. BMJ Open. 2025 Mar 6;15(3):e099414. doi: 10.1136/bmjopen-2025-099414. PMID 40050056

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-01-05): https://cdn.clinicaltrials.gov/large-docs/86/NCT05672186/Prot_SAP_001.pdf
  • Informed Consent Form (2023-01-10): https://cdn.clinicaltrials.gov/large-docs/86/NCT05672186/ICF_002.pdf